CLINICAL TRIAL: NCT00003545
Title: A Phase II Study of 506U78 in Patients With Refractory or Relapsed T-Lineage Acute Lymphoblastic Leukemia (ALL) or Lymphoblastic Lymphomas (LBL)
Brief Title: 506U78 in Treating Patients With Refractory or Relapsed Acute Lymphoblastic Leukemia or Lymphoblastic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01840; CLB-19801; SWOG-C19801; CDR0000066600 (Other Grant/Funding Number: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-02-16 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2007-04

CONDITIONS: Leukemia; Lymphoma
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood lymphoblastic lymphoma; recurrent adult acute lymphoblastic leukemia; T-cell childhood acute lymphoblastic leukemia; T-cell adult acute lymphoblastic leukemia; recurrent adult lymphoblastic lymphoma; recurrent adult T-cell leukemia/lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — nelarabine

ARMS (1):
- Arm I (Experimental): Patients receive 506U78 IV over 2 hours on days 1, 3, and 5. If residual leukemia/lymphoma is present on day 22, then patients receive a second course of 506U78. If day 22 marrow is hypocellular, then a repeat bone marrow biopsy should be obtained on day 29 to assess response. For day 22 or 29 marrow that is in complete response, patients receive 506U78 for two more courses on days 1, 3, and 5, administered every 21 days. Patients are followed every 3 month for 1 year, then every 6 months for a maximum of 10 years.
  Interventions: Drug: nelarabine

INTERVENTIONS:
Drug: nelarabine

SUMMARY:
Phase II trial to study the effectiveness of 506U78 in treating patients with refractory or relapsed acute lymphoblastic leukemia or lymphoblastic lymphoma. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the complete and partial remission rates, as well as the remission duration, in patients with refractory or relapsed T-cell acute lymphoblastic leukemia or lymphoblastic lymphoma receiving 506U78 on an alternate day schedule (days 1, 3, 5).

II. Determine the safety and toxicity of 506U78 administered on this schedule to this patient population.

OUTLINE:

Patients receive 506U78 IV over 2 hours on days 1, 3, and 5. If residual leukemia/lymphoma is present on day 22, then patients receive a second course of 506U78. If day 22 marrow is hypocellular, then a repeat bone marrow biopsy should be obtained on day 29 to assess response. For day 22 or 29 marrow that is in complete response, patients receive 506U78 for two more courses on days 1, 3, and 5, administered every 21 days. Patients are followed every 3 month for 1 year, then every 6 months for a maximum of 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of T-cell acute lymphoblastic leukemia (ALL) or lymphoblastic lymphoma (LBL)
* Leukemia or lymphoma cells should express at least two of the following cell surface antigens: CD1a, CD2, CD3 (surface or cytoplasmic), CD4, CD5, CD7, and CD8
* Leukemia cells should be negative for myeloperoxidase or Sudan Black B If the only T cell markers present are CD4 and CD7, the leukemic cells should be demonstrated to lack the myeloid markers CD33 and/or CD13
* Refractory to at least one induction treatment regimen or in first or later relapse after achieving a complete remission
* No CNS leukemia or lymphoma requiring intrathecal or craniospinal radiotherapy

PATIENT CHARACTERISTICS:

* Age: 16 and over
* Bilirubin no greater than 2 times upper limit of normal (unless due to leukemia)
* Creatinine clearance at least 50 mL/min (unless due to leukemia)
* No neurologic toxicity of grade 3 or greater during prior treatment of ALL/LBL
* No preexisting neuropathy of grade 2 or greater regardless of causality
* No history of seizure disorder
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No concurrent erythropoietin
* No other concurrent chemotherapy
* No concurrent dexamethasone or other steroidal antiemetics
* No concurrent hormone therapy, except for non-disease-related conditions

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 1998-08; Primary Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel DeAngelo, MD, PhD, Study Chair — Dana-Farber Cancer Institute; Steven E. Coutre, MD, Study Chair — Stanford University
Locations (91):
- United States (91):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Stanford University, Stanford, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Cancer Center, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington

REFERENCES:
- [Result] DeAngelo DJ, Yu D, Johnson JL, Coutre SE, Stone RM, Stopeck AT, Gockerman JP, Mitchell BS, Appelbaum FR, Larson RA. Nelarabine induces complete remissions in adults with relapsed or refractory T-lineage acute lymphoblastic leukemia or lymphoblastic lymphoma: Cancer and Leukemia Group B study 19801. Blood. 2007 Jun 15;109(12):5136-42. doi: 10.1182/blood-2006-11-056754. Epub 2007 Mar 7. PMID 17344466
- [Result] De Angelo DJ, Yu D, Dodge RK, et al.: A phase II study of 2-amino-9-b-D-arabinosyl-6-methoxy-9H-purine (506U78) in patients with relapsed or refractory T-Lineage acute lymphoblastic leukemia (ALL) or lymphoblastic lymphoma (LBL): CALGB study 19801. [Abstract] Blood 100 (11 Pt 1): A-743, 2002.